CLINICAL TRIAL: NCT05393401
Title: Photoplethysmographic Measurements of Pulse Wave Velocity (PWV) and Blood Pressure (BP) MEPPAVOP
Brief Title: Photoplethysmographic Measurements of Pulse Wave Velocity (PWV) and Blood Pressure (BP)
Acronym: MEPPAVOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 38RC21.0460
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Photoplethysmography; Pulse Wave Velocity (PWV); Blood Pressure (BP)

STUDY DESIGN:
Intervention Model Description: The Primary Purpose of this clinical trial is to test a prototype device for feasibility and not health outcomes. This study is conducted to confirm the design and operating specifications of a device before beginning a full clinical trial. Primary Purpose is therefore "Device Feasibility"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VOP1k (Experimental): Medical Device
  Interventions: Device: VOP1k

INTERVENTIONS:
Device: VOP1k — Photoplethysmographic records

SUMMARY:
Theoretically, there is a correlation between the PWV and the value of the BP, mediated by the distensibility of the segment of artery where the measurements take place. The hypothesis is therefore that the measurement of the PWV through a multisite medical device for detecting the pulse wave by photoplethysmography makes it possible to deduce the value of the BP.

DETAILED DESCRIPTION:
The aim is to test on healthy volunteers a prototype of a non-invasive, non-CE marked medical device (VOP1k ) for the continuous monitoring of pulse wave velocity (PWV) and to study the relationship between this value and the blood pressure (BP). Indeed, the monitoring of hemodynamic parameters constitutes an essential element of the basal monitoring of patients. Among these parameters, the most used and the most routine is the measurement of BP. This measurement makes it possible in particular to detect the presence or absence of arterial hypertension (HTA), which is a major cause of premature mortality, of high prevalence within the population, involving high medical costs. Contrary to what one might think, the practice of measuring BP is not completely satisfactory, each of the techniques used having characteristics likely to lead to errors of judgment. Oscillometric and auscultatory techniques give discontinuous measurements, expose to the white coat effect when they are performed by a caregiver. Arterial occlusion by external back pressure, which is the basis of these measurement techniques, causes erroneous results and discomfort during repetitive measurements. The use of commercial semi-automatic BP monitors is fraught with validation problems. The necessary confirmation of the diagnosis of hypertension, which is based on ambulatory measurements for 24 hours using these devices, is therefore questionable. The diagnosis of the importance of arterial damage at the base of hypertension could be carried by measurements of the PWV which reflects the stiffness of the arteries. However, this diagnostic means is not currently based on a technology that can be used routinely. Means of measuring BP and arterial stiffness by invasive techniques, which are themselves subject to the risk of poor signal transmission, cannot be used outside the hospital, due to the associated risks. Non-invasive continuous measurement by the volume clamp technique, although devoid of the risks of arterial catheterization, is not available outside specialized hospital departments, and also has the disadvantage of relying on the use of external counter pressure.The technique of measurement by (photoplethysmography (PPG)), i.e. the use of an optical sensor, placed in a non-invasive way on the path of a shallow artery, makes it possible to detect the passage of the pulse wave . The combined use of several sensors located at a distance from each other on the path of the same artery, thus makes it possible to determine the velocity of the pulse wave. This technique can potentially measure over short distances, which limits the sources of error, and allows continuous measurement without discomfort. Moreover, it is compatible with low-cost integration. Indeed, acquisition technologies based on microelectronics are widely developed and mature since their massive use in smartphones. The measurement of PWV makes it possible to quantify arterial stiffness, which is a direct risk factor for morbidity and mortality associated with cardiovascular pathologies. The additional interest of this measurement, in addition to the fact of its non-invasiveness, comes from the fact that there is a correlation between the PWV and the BP, and therefore that the measurement of the PWV can make it possible to obtain a measurement of the BP. It should be noted that one aspect of the aspects of blood pressure measurement consists of being able to measure the central blood pressure, that is to say that which reigns in the aorta. However, most of the measurement techniques used routinely only measure the peripheral arterial pressure, which makes it necessary to use transfer functions to know the central pressure, or to ignore the differences in central pressure/peripheral pressure behavior. The technology proposed for the measurement makes it possible to consider overcoming this problem by placing, in one of the versions, a sensor at the carotid level, which is the arterial segment that best reflects the central pressure, unlike the humeral, femoral or radial segments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy healthy volunteer subject,
* Aged 18 or over,
* Having expressed their consent to the research,
* Affiliated to a social security scheme,
* Registered in the national file of people who lend themselves to biomedical research

Exclusion Criteria:

* People referred to in Articles L1121-5 to L1121-8 of the Public Health Code (corresponds to all protected persons: pregnant, parturient or breastfeeding women, persons deprived of liberty by judicial or administrative decision, persons subject of psychiatric care, minor, and person subject to a legal protection measure: guardianship, curatorship or safeguard of justice)
* Any history or presence of chronic illness
* Presence of Wolf Parkinson White ECG changes
* Subject with orthostatic hypotension
* People with an active implant (e.g. pacemaker)
* Known allergy or intolerance to silicone
* Orthostatic hypotension
* Cutaneous excoriations preventing the placement of sensors on the arms
* Patient with an active implant
* Subject cannot be contacted in case of emergency
* Taking treatment that may impact the recorded physiological measurements
* Subject in period of exclusion from another clinical investigation
* Subject who would receive more than 4500 euros in compensation due to his participation in other biomedical research in the 12 months preceding this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Collect and process the pulse wave signal by the multi-site photoplethysmographic method in order to assess the feasibility and reliability of PWV measurement by this technique in a healthy adult population. | 4 hours
  Measurement of the degree of correlation between the PWV estimated from the device under study and the PWV measured by the "Complior®" reference device. "

SECONDARY OUTCOMES:
Determination of the most adequate distance between the sensors for measuring PWV | 4 hours
  Measurement of the standard PWV deviation measured by the Clearsight device, PWV estimated by the multi-site medical device VOP1k
Study of the relationship between the PWV measured with the device and BP measurement obtained with the gold standard (discrete auscultatory measurements and continuous Clearsight measurements) | 4 hours
  Measurement of the difference between calculated BP and measured brachial BP to check that it does not exceed 5 to 8 mm Hg
Determination of the most adequate algorithm to obtain BP values from PWV | 4 hours
  Calculation of the algorithm to minimize the difference between calculated BP and measured BP
Check that the signal processing makes it possible to adapt to physiological variations in BP in the same individual | 4 hours
  Calculation of the algorithm to minimize the difference between calculated BP and measured BP obtained during PA modifications caused by the different experimental conditions
Check that the signal processing to obtain the BP can be adapted to different individuals | 4 hours
  Calculation of the algorithm to minimize the difference between calculated BP and measured BP

CONTACTS AND LOCATIONS:
Locations (1):
- Clinatec Cea/Chuga, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharman JE, O'Brien E, Alpert B, Schutte AE, Delles C, Hecht Olsen M, Asmar R, Atkins N, Barbosa E, Calhoun D, Campbell NRC, Chalmers J, Benjamin I, Jennings G, Laurent S, Boutouyrie P, Lopez-Jaramillo P, McManus RJ, Mihailidou AS, Ordunez P, Padwal R, Palatini P, Parati G, Poulter N, Rakotz MK, Rosendorff C, Saladini F, Scuteri A, Sebba Barroso W, Cho MC, Sung KC, Townsend RR, Wang JG, Willum Hansen T, Wozniak G, Stergiou G; Lancet Commission on Hypertension Group. Lancet Commission on Hypertension group position statement on the global improvement of accuracy standards for devices that measure blood pressure. J Hypertens. 2020 Jan;38(1):21-29. doi: 10.1097/HJH.0000000000002246. PMID 31790375
- [Background] Vlachopoulos C, Aznaouridis K, O'Rourke MF, Safar ME, Baou K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with central haemodynamics: a systematic review and meta-analysis. Eur Heart J. 2010 Aug;31(15):1865-71. doi: 10.1093/eurheartj/ehq024. Epub 2010 Mar 2. PMID 20197424
- [Background] Bramwell C, Hill and AV, The Velocity of the Pulse Wave in Man, Proc. R. Soc. Lond. B 1922 93, 298-306
- [Background] Lubin M, Vray D, Bonnet S. Blood pressure measurement by coupling an external pressure and photo-plethysmographic signals. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:4996-4999. doi: 10.1109/EMBC44109.2020.9176730. PMID 33019108
- [Background] Block RC, Yavarimanesh M, Natarajan K, Carek A, Mousavi A, Chandrasekhar A, Kim CS, Zhu J, Schifitto G, Mestha LK, Inan OT, Hahn JO, Mukkamala R. Conventional pulse transit times as markers of blood pressure changes in humans. Sci Rep. 2020 Oct 2;10(1):16373. doi: 10.1038/s41598-020-73143-8. PMID 33009445